CLINICAL TRIAL: NCT03072043
Title: A Phase 1b/2 Study to Evaluate the Safety and Efficacy of APR-246 in Combination With Azacitidine for the Treatment of TP53 Mutant Myeloid Neoplasms
Brief Title: Phase 1b/2 Safety and Efficacy of APR-246 w/Azacitidine for tx of TP53 Mutant Myeloid Neoplasms
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18973
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia; Myeloproliferative Neoplasm; Chronic Myelomonocytic Leukemia
Keywords: myelodysplastic syndrome (MDS); TP53 mutant myelodysplastic syndrome; MDS/myeloproliferative neoplasm (MPN); chronic myelomonocytic leukemia (CMML); acute myeloid leukemia (AML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic | interventions — eprenetapopt; Azacitidine

STUDY DESIGN:
Intervention Model Description: Phase 1b Dose Escalation followed by Phase 2 treatment. Participants will be evaluable for inclusion in the Phase 1b and Phase 2 portions of the study if they receive at least one dose of protocol therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b Dose Escalation (Experimental): Participants will receive intravenous infusions of APR-246 as a lead-in phase on days -14 to -11 starting at Dose Level 1 prior to starting cycle #1 of combination therapy with azacitidine. Combination therapy will consist of APR-246 on days 1-4 and azacitidine on days 4-10 (or days 4-5 and 8-12) of a 28 day cycle.
  Interventions: Drug: APR-246; Drug: Azacitidine
- Phase 2 Treatment (Experimental): Participants will be treated with APR-246 administered at the maximum tolerated dose (MTD) with azacitidine on a 28 day cycle utilizing the same dosing schedule as in Phase 1b.
  Interventions: Drug: APR-246; Drug: Azacitidine

INTERVENTIONS:
Drug: APR-246 — Phase 1b: Dose escalation of APR-246 via intravenous (IV) infusion, with starting dose of 50 mg/kg lean body weight (LBW). Phase 2: APR-246 at maximum tolerated dose (MTD).
  Other Names: PRIMA-1MET; Methylated analogue to PRIMA-1
Drug: Azacitidine — Azacitidine is administered subcutaneously (SC) or via IV at 75 mg/m^2.
  Other Names: Mylosar; Vidaza

SUMMARY:
The main purpose of this study is to determine the safe and recommended dose of APR-246 in combination with azacitidine as well as to see if this combination of therapy improves overall survival.

DETAILED DESCRIPTION:
Participants will be treated for a total of 6 cycles. For participants responding or who have stable disease following cycle 6, treatment may continue until one of the following criteria applies:

* Inter-current illness that prevents further administration of treatment,
* Unacceptable adverse event(s),
* Participant decides to withdraw from the study, or
* General or specific changes in the participant's condition render the participant unacceptable for further treatment in the judgment of the investigator.
* Evidence of disease progression by the International Working Group (IWG) 2006 criteria.

Participants who wish not to continue treatment at time of disease assessment at end of cycle 6 will complete their end of treatment visit upon completion of cycle 6.

ELIGIBILITY:
Inclusion Criteria:

* Has signed the Informed Consent (ICF) and is able to comply with protocol requirements.
* Has adequate organ function according to study protocol guidelines.
* Age ≥18 years at the time of signing the informed consent form.
* Documented diagnosis of myelodysplastic syndrome (MDS), MDS/ myeloproliferative neoplasm (MPN), chronic myelomonocytic leukemia (CMML) or oligoblastic AML (20-30% myeloblasts) by World Health Organization (WHO) criteria.
* Documentation of a TP53 gene mutation by NGS based on central or local evaluation.
* For TP53 mutant patients with lower risk MDS (i.e., low or intermediate-1 risk by the International Prognostic Scoring System (IPSS)) and isolated deletion of 5q (del(5q)), failure of prior treatment with at least 4 full cycles of lenalidomide defined as no response to treatment, loss of response at any time point, progressive disease, or intolerance to therapy.
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 is required.
* If of childbearing potential, negative pre-treatment urine or serum pregnancy test.
* If of childbearing potential, willing to use an effective form of contraception such as hormonal birth control, intrauterine device or double barrier method during chemotherapy treatment and for at least six months thereafter.

Exclusion Criteria:

* Known history of HIV or active hepatitis B or active hepatitis C infection (testing not mandatory).
* Has any of the following cardiac abnormalities (as determined by treating MD): a. Symptomatic congestive heart failure; b. Myocardial infarction less than or equal to 6 months prior to enrollment; c. Unstable angina pectoris; d. Serious uncontrolled cardiac arrhythmia; e. QTc ≥ 470 msec
* Concomitant malignancies or previous malignancies with less than a 1-year disease free interval at the time of signing consent. Potential participants with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (e.g., cervix) may enroll irrespective of the time of diagnosis.
* Use of cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of MDS, MDS/MPN, CMML or AML within 14 days of the first day of study drug treatment.
* No concurrent use of erythroid stimulating agents, G-CSF, GM-CSF is allowed during study except in cases of febrile neutropenia where G-CSF can be used for short term. Growth factors must be stopped 14 days prior to study.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sallman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Sallman DA, DeZern AE, Garcia-Manero G, Steensma DP, Roboz GJ, Sekeres MA, Cluzeau T, Sweet KL, McLemore A, McGraw KL, Puskas J, Zhang L, Yao J, Mo Q, Nardelli L, Al Ali NH, Padron E, Korbel G, Attar EC, Kantarjian HM, Lancet JE, Fenaux P, List AF, Komrokji RS. Eprenetapopt (APR-246) and Azacitidine in TP53-Mutant Myelodysplastic Syndromes. J Clin Oncol. 2021 May 10;39(14):1584-1594. doi: 10.1200/JCO.20.02341. Epub 2021 Jan 15. PMID 33449813
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b Dose Level 1: Participants treated at level 1: APR-246 50mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
- Phase 1B Dose Level 2: Participants treated at dose level 2: APR-246 75mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
- Phase 1B Dose Level 3 / Phase 2 MTD: Participants treated at dose level 3/Phase 2 MTD : APR-246 100 mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
Period: Overall Study
Arm/Group | Phase 1b Dose Level 1 | Phase 1B Dose Level 2 | Phase 1B Dose Level 3 / Phase 2 MTD
Started | 3 | 3 | 49
Completed | 3 | 3 | 40
Not Completed | 0 | 0 | 9
Not completed — Death | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Phase 1B Dos Level 2: Participants treated at dose level 2: APR-246 75mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
- Phase 1B Dose Level 3/ MTD: Participants treated at dose level 3/MTD : APR-246 100 mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
- Total: Total of all reporting groups
Arm/Group | Phase 1B Dose Level 1 | Phase 1B Dos Level 2 | Phase 1B Dose Level 3/ MTD | Total
Number analyzed (Participants) | 3 | 3 | 49 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 20 | 22
  >=65 years | 2 | 2 | 29 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 24 | 29
  Male | 1 | 0 | 25 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 1 | 45 | 49
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 2 | 3 | 42 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 49 | 55

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD)
Description: Maximum Tolerated Dose, defined as the dose level below which dose limiting toxicity (DLT) is manifested in ≥33% of the patients or at dose level 3 if DLT is manifested in <33% of the patients.
Time Frame: Up to 12 months
Measure: Number; unit: mg/day
Arm/Group | Phase 1b Dose Escalation
Number analyzed (Participants) | 12
mg/day | 4500

2. Primary Outcome: Phase 2: Complete Response (CR) Rate
Description: Complete Response Rate as defined by the 2006 International Working Group (IWG) criteria.
Time Frame: Up to 12 months
Population: 45 participants were evaluable for response
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Phase 2: Participants in Dose Level 3/MTD: All participants who received at least one dose at level 3: 100 mg/kg LBW APR-246 + 75 mg Azacitidine
Arm/Group | Phase 2: Participants in Dose Level 3/MTD
Number analyzed (Participants) | 45
percentage of patients | 53 [38 to 68]

3. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response defined as the time between achieving response and progression of disease.
Time Frame: Up to 24 months
Population: 45 participants were evaluable for response.
Measure: Median (Full Range); unit: months
Groups:
- Evaluable Participants: All evaluable participants
Arm/Group | Evaluable Participants
Number analyzed (Participants) | 45
months | 8 [6.5 to 11.2]

4. Secondary Outcome: Overall Survival (OS)
Description: OS:The length of time from the start of treatment until death by any cause.
Time Frame: Up to 24 months
Population: All participants who received at least one dose of study drug
Measure: Median (Full Range); unit: months
Groups:
- Phase 1B Dose Level 1: All participants treated at level 1: APR-246 50mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
- Phase 1B Dose Level 2: All participants treated at dose level 2: APR-246 75mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
- Phase 1B: Dose Level 3 / Phase 2 MTD: All participants treated at dose level 3/ Phase 2 MTD : APR-246 100 mg/kg lean body weight (LBW) + Azacitidine 75mg/m^2
Arm/Group | Phase 1B Dose Level 1 | Phase 1B Dose Level 2 | Phase 1B: Dose Level 3 / Phase 2 MTD
Number analyzed (Participants) | 3 | 3 | 49
months | 14.6 [2.4 to 16.0] | 11.6 [6.3 to 13.7] | 10.4 [0.7 to 17.9]

5. Secondary Outcome: Phase 2: Overall Response Rate
Description: Proportion of participants achieving hematological improvement (HI), partial response (PR), complete response (CR), and/or marrow CR (mCR) by the IWG 2006 criteria.
Time Frame: Up to 24 months
Population: 45 participants were evaluable for response
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 45
percent of participants | 87 [73 to 95]

ADVERSE EVENTS:
Time Frame: 2 years, 10 months
Description: All Serious Adverse Events are reported, regardless of causality. Serious Adverse Events were reported during screening period and within 100 days of discontinuation of dosing.
Groups:
- Phase 1b Dose Level 1: All participants treated at dose level 1: APR-246 50 mg/kg lean body weight (LBW) + Azacitidine 75 mg/m^2
- Phase 1B Dose Level 2: All participants treated at dose level 2: APR-246 75 mg/kg lean body weight (LBW) + Azacitidine 75 mg/m^2
- Phase 1B Dose Level 3/Phase 2 MTD: All participants treated at dose level 3 & Phase 2: APR-246 100 mg/kg lean body weight (LBW) + Azacitidine 75 mg/m^2
Arm/Group | Phase 1b Dose Level 1 | Phase 1B Dose Level 2 | Phase 1B Dose Level 3/Phase 2 MTD
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 36/49
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 30/49
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Dose Level 1 (N=3) | Phase 1B Dose Level 2 (N=3) | Phase 1B Dose Level 3/Phase 2 MTD (N=49)
Blood and Lymphatic system disorders -Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Escherichia coli
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 17 (34)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain -cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ear and labyrinth disorders -Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Diverticulitis
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi organ failure (General disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection and Infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 7 (9)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 7 (7)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5)
Skin inefection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Vascular disorders -Other (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) — Deep vein thrombosis
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Diffuse body pain
Vascular disorders - Other (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — subdural hematoma
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Dose Level 1 (N=3) | Phase 1B Dose Level 2 (N=3) | Phase 1B Dose Level 3/Phase 2 MTD (N=49)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (8) | 32 (57)
Blurry vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 12 (16)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 7 (18)
Generalized edema (General disorders) | 1 (1) | 0 (0) | 1 (4)
Pain -Side pain (General disorders) | 0 (0) | 0 (0) | 2 (2) — Generalized right side pain
Pain -Hip (General disorders) | 1 (1) | 0 (0) | 4 (4) — Hip pain
Pain- Jaw (General disorders) | 0 (0) | 1 (1) | 0 (0) — Jaw pain
Pain -Shoulder (General disorders) | 0 (0) | 0 (0) | 4 (4) — Shoulder pain
Pain -Muscle (General disorders) | 0 (0) | 0 (0) | 1 (1) — muscle pain
Pain -Chest (General disorders) | 0 (0) | 0 (0) | 1 (1) — Heartburn
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — Hepatomegaly
Port vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Allergic reaction including pruritis (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Allergic Reaction - swollen tongue (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Swollen tongue related to urinary tract infection medication
Infections and Infestations - Other (Infections and infestations) | 3 (3) | 1 (4) | 12 (17)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Rhinitis, infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 7 (8)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Heart palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders -Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — Ringing in ears
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 2 (2) — Stye in eye
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 21 (24)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 15 (24)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (10)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (5) | 22 (37)
Edema- limbs (General disorders) | 0 (0) | 0 (0) | 18 (21)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (2) — Platelet transfusion reaction
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Investigations) | 2 (5) | 2 (7) | 12 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 9 (10)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 8 (14)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 4 (11)
Dizziness (Nervous system disorders) | 1 (1) | 2 (5) | 18 (31)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (8) | 12 (13) — facial numbness
Headache (Nervous system disorders) | 1 (2) | 1 (2) | 14 (16)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 10 (21)
Chills (General disorders) | 0 (0) | 0 (0) | 8 (9)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 6 (7)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 14 (19)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 10 (14)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 6 (11)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 8 (13)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (4) | 3 (12) | 10 (27)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 14 (15)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Investigations) | 1 (1) | 0 (0) | 7 (11)
Hypomagnesemia (Investigations) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (8)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 10 (14)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (7)
Allodynia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (6)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 5 (6)
Nervous system disorders -Other (Nervous system disorders) | 0 (0) | 0 (0) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Injury, poisoning and procedural complications - other (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 4 (5)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 23 (38)
Brusing (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Cecal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Dental carries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 16 (17)
Edema face (General disorders) | 0 (0) | 0 (0) | 2 (2)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders -other (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (3) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (4)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 12 (12)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (6) | 12 (23)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Palmar-plantar ethryodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (9)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness - lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6)
Malaise (General disorders) | 0 (0) | 0 (0) | 3 (4)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 1 (3)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (8)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (6)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diffuse body pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03072043/Prot_SAP_000.pdf